CLINICAL TRIAL: NCT06171971
Title: Evaluation of the Clinical and Therapeutic Impact of Large Genomic Studies at Diagnosis in Pediatric Solid Cancers
Brief Title: Clinical and Therapeutic Impact of Large Genomic Studies at Diagnosis in Pediatric Solid Cancers
Acronym: CS-PEDIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8661
Record Dates: First submitted 2022-09-06; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Pediatric Solid Tumors
Keywords: Pediatric solid tumors; BROAD GENOMIC STUDIES; SOLID CANCERS; Genomic medicine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pediatric solid tumors with an unfavorable prognosis remain a public health issue due to their morbidity and mortality and their rapidly evolving profile. They are defined by an expected overall survival of < 30%. Progress has been made in genomic medicine with existing recommendations for the adult population, with the objective of personalized medicine. Recommendations for the pediatric population are still under consideration

ELIGIBILITY:
Inclusion criteria

* Patients of pediatric age up to 22 years included at the time of molecular analysis
* Histological carcinological diagnosis performed at HUS
* Carcinological follow-up performed at HUS
* Patients with a solid tumor of unfavorable prognosis, refractory or in relapse
* Molecular analysis performed on tumor or blood samples
* Adult patients who do not object to the re-use of their personal data for medical research purposes
* Minor patients and their parents who do not object to the re-use of their personal data for scientific research purposes.

Criteria for non-inclusion

* Molecular biology results not usable due to poor sample quality or insufficient genetic material
* Patients who have expressed their opposition to participate in the study
* Parental authority holders who have expressed their opposition to participate in the study

Ages: 1 Year to 22 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients of pediatric age up to 22 years included at the time of molecular analysis
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Retrospective description of the clinical and therapeutic impact of the systematic performance of molecular analyzes on solid tumors | up to 12 months
  The aim of this retrospective study is to improve and harmonize international practices

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'onco-hématologie pédiatrique - CHU de Strasbourg - France, Strasbourg, France